CLINICAL TRIAL: NCT05040711
Title: Piloting an mHealth-delivered Mindfulness Therapy With Patients With Serious Illness and Their Caregivers to Alleviate Symptoms of Anxiety
Brief Title: mHealth Mindfulness With Patients With Serious Illness and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Elissa Kozlov, Ph.D, Instructor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2021001219
Record Dates: First submitted 2021-09-07; First posted 2021-09-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Caregiver Stress Syndrome; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness coach (Experimental): Mindfulness coach is an app that provides a training plan with 14 sequential levels, a "practice now" area with evidence-based mindfulness audio exercises, assessments using the Five-Factor Mindfulness Questionnaire Short Form (FFMQ-SF)90, and education about mindfulness an iOS- and Android-based app designed to deliver a mindfulness training course centered on Veteran's Affairs (VA) protocols. Developed by the VA's National Center for PTSD, the app provides an engaging introduction to MT, regardless of specific psychiatric illness or patient population. . To progress to the next level, the user must interact with every element. The training plan levels include psychoeducation and exercises (guided meditations and seated practices), which increase in duration as users progress. Levels 1,7 and 14 also include an assessment with the FFMQ-SF. The "practice now" area has guided meditations to practice new skills.
  Interventions: Behavioral: Mindfulness Coach
- control - web MD (Active Comparator): A a widely available health and wellness app that provides users with daily content on general health, WebMD, will serve as the attention control. Similar health-based apps have been used as controls in other mHealth psychotherapy intervention trials.100,101 The control group will be instructed to access the app 4x/week (same as intervention group) and will receive an orientation and 2 booster sessions as well. I considered other control group options including treatment as usual, but attention control was selected due to the variability of treatment as usual.
  Interventions: Behavioral: Active Comparator

INTERVENTIONS:
Behavioral: Mindfulness Coach — This study will use Mindfulness Coach, an iOS- and Android-based app designed to deliver a mindfulness training course centered on Veteran's Affairs (VA) protocols. Developed by the VA's National Center for PTSD, the app provides an engaging introduction to MT, regardless of specific psychiatric illness or patient population. The app provides a training plan with 14 sequential levels, a "practice now" area with evidence-based mindfulness audio exercises, assessments using the Five-Factor Mindfulness Questionnaire Short Form (FFMQ-SF)90, and education about mindfulness. To progress to the next level, the user must interact with every element. The training plan levels include psychoeducation and exercises (guided meditations and seated practices), which increase in duration as users progress. Levels 1,7 and 14 also include an assessment with the FFMQ-SF. The "practice now" area has guided meditations to practice new skills.
  Arms: mindfulness coach
Behavioral: Active Comparator — A a widely available health and wellness app that provides users with daily content on general health, WebMD, will serve as the attention control. Similar health-based apps have been used as controls in other mHealth psychotherapy intervention trials.100,101 The control group will be instructed to access the app 4x/week (same as intervention group) and will receive an orientation and 2 booster sessions as well. I considered other control group options including treatment as usual, but attention control was selected due to the variability of treatment as usual.
  Other Names: WebMD
  Arms: control - web MD

SUMMARY:
Older adults with serious illness and their caregivers have high rates of anxiety and limited access to effective, non-pharmacological treatments. A recent National Academy of Medicine report recommended increased emphasis on disseminating and implementing evidence-based psychotherapies in order to have maximal public health impact. Through this work, I will identify a sustainable and potentially scalable dyadic intervention and delivery model to manage symptoms of anxiety in older adults with serious illness and their caregivers in primary care.

DETAILED DESCRIPTION:
Research: Up to 70% of adults with serious illness have symptoms of anxiety. Undiagnosed and undertreated anxiety contributes to higher risk of pain, depression, fatigue, dyspnea, and polypharmacy. Patients with high symptom burden and anxiety heavily impact family caregivers, which nearly 8 million older adults in the U.S. rely on for assistance. Decades of research reveal the negative effects of caregiving on caregivers, (e.g., high levels of stress, depression, and anxiety). Furthermore, there is a mutuality of distress in the caregiver/patient dyad - when patients suffer psychologically, the caregiver suffers too. Unfortunately, older adults and their caregivers have limited access to mental health resources because of shortages of mental health providers as well as logistical issues including time constraints, transportation, and scheduling. The objective of this study is to evaluate the feasibility, acceptability, and preliminary efficacy of Mindfulness Coach, an mHealth Mindfulness Therapy intervention developed by the Veterans Affairs, to reduce anxiety in older adults with serious illness and their family caregivers. An efficacious and scalable behavioral intervention that mitigates symptoms of patient and caregiver anxiety has the potential to reduce distress and enhance coping in the patient-caregiver dyad without contributing to polypharmacy or burdensome appointments. Research is urgently needed to evaluate the feasibility, acceptability, and preliminary efficacy of dyadic mHealth mindfulness therapy in older adults with serious illness and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* adults 60+
* Diagnosis of or caregiver for individual with serious illnesses (e.g., ESRD, Cancer, CHF, COPD, Liver Disease)
* Hads-A > 8 for patient or caregiver
* Blessed<6
* fluent in English
* vision and hearing does not interfere with mobile device use
* caregivers who must be 21+
* caregiver must identify as primary source of informal care for patient
* Caregiver blessed <6
* caregiver is fluent in English
* Caregiver's vision and hearing does not interfere with mobile device use.

Exclusion Criteria:

* experience with mindfulness therapy in last 2 years
* not fluent in English
* vision or hearing that impairs use of mobile device
* cognitive impairment more than 6 on Blessed.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale - Anxiety Sub Scale | 6 months
  Anxiety scale with range from 0-21 with higher scores denoting highest anxiety
Hospital Anxiety and Depression Scale - Anxiety Sub Scale | 8 weeks
  Anxiety scale with range from 0-21 with higher scores denoting highest anxiety

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale - Depression Sub Scale | 6 months
  Depression scale with range from 0-21 with higher scores denoting highest depression
Hospital Anxiety and Depression Scale - Depression Sub Scale | 8 weeks
  Depression scale with range from 0-21 with higher scores denoting highest depression
Perceived stress scale | 8 weeks
  Scale with range from 0 - 40 with higher values indicating more perceived stress

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Kozlov, PhD, Principal Investigator — Rutgers University
Locations (3):
- United States (3):
  - RWJ Barnabas Outpatient Geriatric Clinics, Livingston, New Jersey
  - RWJB Outpatient Geriatrics, Monroe, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No